CLINICAL TRIAL: NCT03825887
Title: Evaluation of Safety and Efficacy of Nalbuphine Versus Morphine Patient Controlled Analgesia (PCA) for Mucositis Pain in Pediatric Patients. A Prospective Randomized Double Blinded Clinical Trial
Brief Title: Nalbuphine Versus Morphine for Mucositis Pain in Pediatric Cancer Patients
Acronym: PCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CCHE -BM0001
Record Dates: First submitted 2019-01-22; First posted 2019-01-31 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-07

CONDITIONS: Acute Myeloid Leukemia; Stem Cell Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute | interventions — Nalbuphine; Morphine

STUDY DESIGN:
Intervention Model Description: patients with AML , ALL and bone marrow transplantation with oral mucositis grade3 or 4 were randomized into two group: patient using of PCA Morphine (Group A) patient using of PCA Nalbuphine (Group B). Patients of both groups will be started on the same dose of 10 mcg / kg / hour as a background and 10 mcg bolus dose with lock-out 20 minutes having the maximum allowed dose up to 40 mcg / hour.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A-PCA Morphine (Active Comparator): Patients will be started on the same dose of 10 mcg / kg / hour as a background and 10 mcg bolus dose with lock-out 20 minutes having the maximum allowed dose up to 40 mcg /kg/ hour.
  Interventions: Drug: Morphine
- Group B-PCA Nalbuphine (Experimental): Patients will be started on the same dose of 10 mcg / kg / hour as a background and 10 mcg bolus dose with lock-out 20 minutes having the maximum allowed dose up to 40 mcg /kg/ hour.
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Nalbuphine — Nalbuphine (Group B): Patients will be started on the same dose of 10 mcg / kg / hour as a background and 10mcg bolus dose with lock-out 20 minutes having the maximum allowed dose up to 40mcg /kg/ hour.
  Any patient will continue to complain of pain rating 4-6 on VAS after reaching the maximum designated dose (which is 40 mcg/kg/hour) will be transferred to the ICU for close monitoring according to the internal hospital guidelines and getting him/her out of the study.
  There is no drug shifting at any part of the study.
  Arms: Group B-PCA Nalbuphine
Drug: Morphine — morphine (Group A): Patients will be started on the same dose of 10 mcg / kg / hour as a background and 10mcg bolus dose with lock-out 20 minutes having the maximum allowed dose up to 40mcg /kg/ hour.
  Any patient will continue to complain of pain rating 4-6 on VAS after reaching the maximum designated dose (which is 40 mcg/kg/hour) will be transferred to the ICU for close monitoring according to the internal hospital guidelines and getting him/her out of the study.
  There is no drug shifting at any part of the study.
  Arms: Group A-PCA Morphine

SUMMARY:
Evaluation of safety and efficacy of Nalbuphine versus Morphine patient controlled analgesia (PCA) for mucositis pain in pediatric cancer patients

DETAILED DESCRIPTION:
The investigators will compare between using of PCA Morphine (Group A) and using of PCA Nalbuphine (Group B) in the following items over the first 7 days of initiation:

1. Pain intensity VAS every 12 hours and during the performing of mouth care for each patient over the first 7 days.
2. Total opioid consumptions for each patient every 24 hours and the total consumption of the entire 7 days since initiation.
3. Number of active and total pushes of PCA buttons every 24 hours and the sum up of the active and total pushes of PCA buttons for each patient over the 7 days.
4. Patient satisfaction at the end of the 7 days. Patient satisfaction score PSS was assessed using a linear scale where 0=very satisfied; 10=very dissatisfied (14).
5. Serious adverse events. (Nausea and vomiting, pruritus, respiratory depression, urinary retention, sedation, bradycardia, hypotension).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Primary AML or HSCT and ALL with oral mucositis grade III OR IV presenting in the study period.
* Age above 5 year and below 18 years
* Written Informed Consent from parents/guardian

Exclusion Criteria:

* History of mental retardation
* known or suspected allergy to any narcotics
* Presence of any other co-morbidity:
* kidney (Crcl <50)
* liver (liver enzymes more than 10 folds)
* chest (SPO2 <92% on room air)
* cardiac disease (ejection fraction <40%)
* terminal patients who scheduled for palliative care

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
measure the change in Pain intensity | change occur every 12 hours and during the performing of mouth care for each patient over the first 7 days
  change in pain intensity by visual analogue scale (scale from 0 to 100)
Total opioid consumptions | the total consumption through the entire 7 days since initiation
  total dosing in mg/day

SECONDARY OUTCOMES:
Number of active and total pushes of PCA buttons | every 24 hours and the sum up of the active and total pushes of PCA buttons for each patient over the 7 days.
  Number of active and total pushes of PCA buttons
Patient satisfaction: linear scale | at the end of the 7 days.
  Patient satisfaction score PSS was assessed using a linear scale where 0=very satisfied; 10=very dissatisfied (14).
Assess serious adverse events | during 7 days of treatment only
  by reporting the number of patients with Nausea and vomiting and/or pruritus and/or respiratory depression and/or urinary retention and/or sedation and/or bradycardia and/or hypotension).

CONTACTS AND LOCATIONS:
Locations (1):
- CCHE, Cairo, Egypt